CLINICAL TRIAL: NCT06289127
Title: Test Properties of Lower Quarter Y-Balance Test: Effect of Verbal Instructions and Focus Techniques
Status: Completed | Type: Observational
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Elif Turgut, Associate Professor Elif TURGUT, Hacettepe University
Other Study IDs: GO 22/595
Record Dates: First submitted 2024-02-23; First posted 2024-03-01 (Actual); Last update posted 2024-03-04 (Actual); Status verified 2024-03

CONDITIONS: Healthy; Attention Disturbances; Physical Stress
Keywords: Balance; Focus techniques; Performance; Verbal instructions

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: Lower Quarter Y Balance Test — The LQYBT is a widely used test for assessing lower extremity dynamic balance and neuromuscular control. Participants' lower limb balance was performed using The Y Balance Test Kit™ (Move2Perform, Evansville, IN).

SUMMARY:
The Lower Quadrant Y-Balance Test (LQYBT) is a landmark test used in assessing lower extremity performance, determining risk factors for injury, and making return-to-sport decisions. Studies have shown that the individual's focus of attention affects balance. The literature, has shown that the use of external focus is more effective than the use of internal focus in the execution of a movement.Consistent with these findings, the use of an external focus instruction during the LQYBT may lead to achieve more realistic and a higher performance outcome than the test result with standard instructions. The primary aim of this study was to investigate the effects of using different instructions and focusing techniques on test performance on the LQYBT. The secondary aim was to investigate the reliability of the different instructions and focus tests we used for the LQYBT.

Hypothesis of the study that test performance can be further enhanced by differentiating the instructions and focus techniques. A more effective assessment of individual performance may help us to make a more realistic decision to return to sport.

DETAILED DESCRIPTION:
This study is a prospective cross-sectional research. A total of 52 healthy individuals participated in this study. The test protocols were compeleted in two sessions for each participant. In the first session, participants whose eligibility for the study was determined, were recorded demographic data including age, height, body weight, body mass index, lower extremity dominance, and leg length. Subsequently, the Lower Quarter Y Balance Test (LQYBT) was conducted using three different focus instructions: (1) standardized instruction, (2) internal focus instruction, (3) external focus instruction. Each focus instruction was sequentially applied three times in each direction. The three different instructions were randomized and performed in a different sequence for each participant. In second session, to assess the test-retest reliability of different focus instructions during test, the LQYBT was repeated under the same conditions three days later, by the same researcher.

To ensure normalization, the average distances measured in the anterior, posteromedial, and posterolateral directions were obtained for each command, and the results were divided by the length of the leg and multiplied by 100. The total score for the dominant side in the LQYBT was determined by aggregating the average reach distance across three directions, dividing it by three times the length of the leg, and then multiplying by 100.

ELIGIBILITY:
Inclusion Criteria:

* 18-35 years,
* Currently without pain in lower extremity,
* No history of lower extremity musculoskeletal problems or surgery in the last 12 months.

Exclusion Criteria:

* Had neurological, systemic, or autoimmune disorders.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy individuals
Sampling Method: Probability Sample
Enrollment: 2 (Actual)
Dates: Start 2022-07-20 (Actual); Primary Completion 2023-02-02 (Actual); Study Completion 2023-11-10 (Actual)

PRIMARY OUTCOMES:
Investigate the effects of using different instructions and focusing techniques on test performance on the LQYBT. | 40 minutes for each participant
  To ensure normalization, the average distances measured in the anterior, posteromedial, and posterolateral directions were obtained for each command, and the results were divided by the length of the leg and multiplied by 100. The total score for the dominant side in the LQYBT was determined by aggregating the average reach distance (cm) across three directions, dividing it by three times the length of the leg, and then multiplying by 100. Repeated Measures Analysis of Variance (ANOVA) was used to analyze comparisons of different instruction.

SECONDARY OUTCOMES:
Investigate the reliability of the different instructions and focus tests we used for the LQYBT. | Performed 2 times in 3 days apart, 40 minutes for each participant
  To determine the test-retest reliability of the test results during different focus instructions, we computed the intraclass correlation coefficients (ICCs) along with corresponding 95% confidence intervals (CIs) between the scores of the first and second results of LQYBT. The ICC value was interpreted as follows: below 0.20 indicates poor reliability; between 0.40 and 0.59 suggests satisfactory reliability; between 0.60 and 0.79 indicates very good reliability; and above 0.80 suggests excellent reliability.

CONTACTS AND LOCATIONS:
Locations (1):
- Hacettepe University, Ankara, Sıhhıye, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No